CLINICAL TRIAL: NCT03260296
Title: Smartphones Addiction and Its Correlations Among Assiut University Students
Brief Title: Smartphones Addiction in Assiut University Students
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mariam Gamal, principle investigator, Assiut University
Other Study IDs: 7990
Record Dates: First submitted 2017-08-20; First posted 2017-08-24 (Actual); Last update posted 2017-08-24 (Actual); Status verified 2017-08

CONDITIONS: Behavior Problem; Addiction
Keywords: smartphones addiction
MeSH Terms: conditions — Mental Disorders; Behavior, Addictive

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- University students: university students who use smartphones
  Interventions: Other: self-administered structured questionnaire

INTERVENTIONS:
Other: self-administered structured questionnaire — Data will be collected by self-administered structured questionnaire. The aim of the study and the way of filling the questionnaire will be explained to the students, and then he/she fills the questionnaire by him/her self.
  The questionnaire will assess smartphones addiction and some of its associated factors and its health consequences

SUMMARY:
Smartphones have become a part of our daily life, the number of people using smartphones is increasing day after day. Easy access to internet is the main advantage of smartphones in comparison to traditional mobile phones, so they are considered as handheld convenient substitutes to computers. People use smartphones for many different purposes such as communication, entertainment, browsing for information, education or business facilitation. Unfortunately the excessive use of smartphones makes people 'addicted' to that type of technology. Past research has shown that older people have less positive attitudes towards a variety of technologies and they are less likely than younger people to embrace new technology, so It seems that the problem of smartphones addiction is most likely to affect young people who are fascinated with new technologies.

DETAILED DESCRIPTION:
What is smartphones addiction? The concept of smartphones addiction is not proposed yet for inclusion in the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-5) as non-substance-related disorder but it can be considered one type of technological addictions which were operationally defined by Griffiths as non-chemical (behavioral) addictions which involve human-machine interaction and usually contain inducing and reinforcing features which may contribute to the promotion of addictive tendencies.

Furthermore, Recent work by Lin, et al identified the criteria for diagnosis smartphones addiction as following:

A. Behavioral criteria (3 or more should be present):

1. Preoccupation with smartphone use, and hence keeping smartphone available all day
2. Recurrent failure to resist the impulse to use the smartphone
3. Tolerance: a markedly increase in the duration of smartphone use is needed to achieve satisfaction
4. Withdrawal: as manifested by a dysphoric mood, anxiety and/or irritability after a period without smartphone use
5. Smartphone use for a period longer than intended
6. Persistent desire and/or unsuccessful attempts to cut down or reduce smartphone use
7. Excessive smartphone use and/or time spent on leaving the use
8. Continued excessive smartphone use despite knowledge of having a persistent or recurrent physical or psychological problems caused by smartphone use

B. Functional impairment criteria (2 or more criteria should be present):

1. Excessive use resulting in persistent or recurrent physical or psychological problems
2. Use in a physically hazardous situations (such as while driving or crossing the street) or situations that have other negative impacts on daily life
3. Use that impairs social relationships or performance at school or work
4. Use that is very time-consuming or causes significant distress C. Exclusion criteria Addictive behavior is not associated with obsessive-compulsive disorder or bipolar disorder

Factors associated with smartphones addiction:

* There are many psychological factors related to smartphones addiction such as anxiety, stress, poor social and family relationship, depression, loneliness, shyness, degree of self-esteem and satisfaction with life.
* Studies have also shown the adverse effects of smartphones addiction on quality of sleep, physical activity and academic performance.
* Smartphones addiction also have harmful physical consequences like headache, blurred vision, neck and shoulder pain and impairment of hand function.

Size of problem:

Prevalence of smartphones addiction in young people varies among countries as shown by studies: 29.6% in Saudi Arabia, 44.6% in Lebanon,16.9% in Switzerland, 21.3% in China and 31.33% in India.

-there is no available data about the size of this of this problem in Egypt so investigators need to conduct this study to determine the prevalence of smartphones addiction among young people and it adverse effect on different aspects.

ELIGIBILITY:
Inclusion Criteria:

* -Egyptian students
* Students in one selected academic year
* Students have smartphones

Exclusion Criteria:

* -Non-Egyptian students
* Students in academic years other than the selected one
* Students having traditional mobile phones or not having mobile phones at all

Ages: 17 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Egyptian Students of Assiut University will be the target population Target students will be selected randomly by using a multistage stratified cluster sampling technique.
  At the first stage, Faculties within Assiut University will be stratified into 3 strata; Practical , Theoretical and Medical then faculties will be chosen randomly from each stratum to end up with 4 faculties (2 theoretical, 1 practical and 1 medical).
  In the second stage, cluster sample will be chosen from one academic year within each faculty (practical sections or small classes). The clusters will be chosen through simple random sample.
Sampling Method: Probability Sample
Enrollment: 693 (Estimated)
Dates: Start 2018-10 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Smartphones addiction scale (SAS) | 6 months
  Prevalence of smartphones addiction and its adverse effects will be evaluated by a self-administered questionnaire guided by smartphones addiction scale developed by Kwon et al.

SECONDARY OUTCOMES:
Factors associated with smartphones addiction questionnaire | 6 months
  the study will assess some associated factors that may be risk factors to smartphones addiction as depression and loneliness

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Lin YH, Lin YC, Lee YH, Lin PH, Lin SH, Chang LR, Tseng HW, Yen LY, Yang CC, Kuo TB. Time distortion associated with smartphone addiction: Identifying smartphone addiction via a mobile application (App). J Psychiatr Res. 2015 Jun;65:139-45. doi: 10.1016/j.jpsychires.2015.04.003. Epub 2015 Apr 10. PMID 25935253
- [Result] Griffiths M. Gambling on the internet: A brief note. J Gambl Stud. 1996 Dec;12(4):471-3. doi: 10.1007/BF01539190. No abstract available. PMID 24234164
- [Result] Demirci K, Akgonul M, Akpinar A. Relationship of smartphone use severity with sleep quality, depression, and anxiety in university students. J Behav Addict. 2015 Jun;4(2):85-92. doi: 10.1556/2006.4.2015.010. PMID 26132913
- [Result] Kim SE, Kim JW, Jee YS. Relationship between smartphone addiction and physical activity in Chinese international students in Korea. J Behav Addict. 2015 Sep;4(3):200-5. doi: 10.1556/2006.4.2015.028. PMID 26551911
- [Result] Kim HJ; DH; Kim JS. The relationship between smartphone use and subjective musculoskeletal symptoms and university students. J Phys Ther Sci. 2015 Mar;27(3):575-9. doi: 10.1589/jpts.27.575. Epub 2015 Mar 31. PMID 25931684
- [Result] Haug S, Castro RP, Kwon M, Filler A, Kowatsch T, Schaub MP. Smartphone use and smartphone addiction among young people in Switzerland. J Behav Addict. 2015 Dec;4(4):299-307. doi: 10.1556/2006.4.2015.037. PMID 26690625
- [Result] Nikhita CS, Jadhav PR, Ajinkya SA. Prevalence of Mobile Phone Dependence in Secondary School Adolescents. J Clin Diagn Res. 2015 Nov;9(11):VC06-VC09. doi: 10.7860/JCDR/2015/14396.6803. Epub 2015 Nov 1. PMID 26672469
- [Result] Long J, Liu TQ, Liao YH, Qi C, He HY, Chen SB, Billieux J. Prevalence and correlates of problematic smartphone use in a large random sample of Chinese undergraduates. BMC Psychiatry. 2016 Nov 17;16(1):408. doi: 10.1186/s12888-016-1083-3. PMID 27855666
- [Result] Kwon M, Lee JY, Won WY, Park JW, Min JA, Hahn C, Gu X, Choi JH, Kim DJ. Development and validation of a smartphone addiction scale (SAS). PLoS One. 2013;8(2):e56936. doi: 10.1371/journal.pone.0056936. Epub 2013 Feb 27. PMID 23468893